CLINICAL TRIAL: NCT00004050
Title: Phase II Study Evaluating the Safety and Efficacy of Neoadjuvant Leuvectin Immunotherapy for the Treatment of Prostate Cancer
Brief Title: Leuvectin Followed By Surgery in Treating Patients With Stage II or Stage III Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Development in prostate cancer indication halted
Sponsor: Vical (Industry)
Collaborators: Jonsson Comprehensive Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCL-1102-202; UCLA-9901077-03B (Other: UCLA); CDR0000067244 (Registry Identifier: PDQ (Physician Data Query)); NCI-G99-1568 (Other: NCI)
Record Dates: First submitted 1999-12-10; First posted 2003-10-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuvectin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Leuvectin (Experimental): 2 intratumoral injections of 1000 ug of Leuvectin
  Interventions: Biological: Leuvectin

INTERVENTIONS:
Biological: Leuvectin — Leuvectin injected intratumorally followed by prostatectomy
  Other Names: Interleukin-2 (IL-2) plasmid DNA/lipid complex

SUMMARY:
RATIONALE: Inserting the gene for interleukin-2 into a person's cancer cells may improve the body's ability to fight cancer. Using Leuvectin to deliver this gene may be an effective treatment for prostate cancer.

PURPOSE: Phase II trial to study the effectiveness of Leuvectin followed by surgery in treating patients who have stage II or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the toxicity and tolerability of neoadjuvant Leuvectin in patients with stage II or III prostate cancer.
* Evaluate the efficacy of this regimen in preventing or delaying manifestations of disease progression as demonstrated by biochemical failure or clinical recurrence in this patient population.

OUTLINE: This is a multicenter study.

Patients receive Leuvectin intraprostatically over 10-30 seconds under ultrasound guidance on day 0 followed by a second injection between days 4 and 7. Between days 8 and 14, patients undergo retropubic prostatectomy.

All patients are followed at 2 months. Patients with a PSA no greater than 0.2 ng/mL are followed at 4 months and 6 months, every 3 months for 12 months, and then every 6 months for 3.5 years in the absence of disease progression or biochemical failure.

ACTUAL ACCRUAL: 13 patients were accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage II or III organ confined prostate cancer

  * Resectable disease (candidate for retropubic prostatectomy)
* Gleason score at least 6
* Prostate specific antigen value (PSA) at least 5 ng/mL
* No significant central nervous system (CNS) disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 80-100%
* Eastern Cooperative Oncology Group (ECOG) 0-1

Life expectancy

* Not specified

Hematopoietic

* White blood cell count (WBC) greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 9.0 g/dL

Hepatic

* Bilirubin normal; serum glutamic oxaloacetic transaminase (SGOT), serum glutamic-pyruvic transaminase (SGPT) less than 3 times upper limit of normal
* Prothrombin time (PT)/partial thromboplastin time (PTT) normal
* Albumin greater than 3.0 g/dL
* Hepatitis B surface antigen negative

Renal

* Creatinine normal

Cardiovascular

* No uncontrolled hypertension
* No significant cardiovascular disease
* No history of ventricular dysfunction or arrhythmia
* No congestive heart failure
* No symptoms of coronary artery disease
* No prior myocardial infarction

Other

* No active autoimmune disease
* No active infection requiring parenteral antibiotics
* HIV negative
* No significant psychiatric disorder that would preclude compliance
* No other malignancy within the past 5 years except curatively treated basal or squamous cell skin cancer
* No diabetes mellitus
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for prostate cancer
* At least 5 years since other prior chemotherapy

Endocrine therapy

* No prior glucocorticoids for prostate cancer
* At least 5 years since other prior glucocorticoids

Radiotherapy

* No prior radiotherapy for prostate cancer
* At least 5 years since other prior radiotherapy

Surgery

* See Disease Characteristics
* At least 4 weeks since prior intrathoracic or intrabdominal surgery
* At least 2 weeks since other major surgery

Other

* At least 10 days since prior anticoagulants or nonsteroidal antiinflammatory agents
* No other neoadjuvant or concurrent anticancer drugs
* No concurrent immunosuppressive drugs
* No other concurrent experimental therapy
* No concurrent parenteral antibiotics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1999-06; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Disease recurrence | 2 years
  Measure timing and rate of disease recurrence

SECONDARY OUTCOMES:
Safety of Leuvectin

CONTACTS AND LOCATIONS:
Overall Officials: Arie Belldegrun, MD, FACS, Study Chair — Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio